CLINICAL TRIAL: NCT02029274
Title: A Double Blind, Randomized, Placebo-controlled Study to Evaluate, Safety, Tolerability, Efficacy and Preliminary Dose-response of BAF312 in Patients With Active Dermatomyositis (DM)
Brief Title: Safety and Efficacy of BAF312 in Dermatomyositis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated prematurely after an interim analysis for futility. The study did not provide any evidence for efficacy of BAF312 in dermatomyositis.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CBAF312X2206; 2013-001799-39 (EudraCT Number)
Record Dates: First submitted 2013-12-02; First posted 2014-01-07 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2018-12

CONDITIONS: Active Dermatomyositis
Keywords: Dermatomyositis
MeSH Terms: conditions — Dermatomyositis | interventions — siponimod

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- BAF312 0.5mg (Experimental): During period 1, participants were uptitrated daily from BAF312 0.25 mg to 0.5 mg over a 10 day period. After, participants continued on 0.5 mg daily for up to 24 weeks. During period 2, participants were uptitrated daily from BAF312 0.25 mg to 2.0 mg over a 10 day period. After, participants continued on 2.0 mg daily for up to 24 weeks.
  Interventions: Drug: BAF312
- BAF312 2mg (Experimental): During period 1, participants were uptitrated daily from BAF312 0.25 mg to 2.0 mg over a 10 day period. After, participants continued on 2.0 mg daily for up to 24 weeks. During period 2, participants were uptitrated daily from BAF312 0.25 mg to 2.0 mg over a 10 day period. After, participants continued on 2.0 mg daily for up to 24 weeks.
  Interventions: Drug: BAF312
- BAF312 10 mg (Experimental): During period 1, participants were uptitrated daily from BAF312 0.25 mg to 10.0 mg over a 10 day period. After, participants continued on 10.0 mg daily for up to 24 weeks. During period 2, participants were uptitrated daily from BAF312 0.25 mg to 2.0 mg over a 10 day period. After, participants continued on 2.0 mg daily for up to 24 weeks.
  Interventions: Drug: BAF312
- Placebo (Placebo Comparator): During period 1, participants received matching placebo daily for up to 24 weeks. During period 2, participants were uptitrated daily from BAF312 0.25 mg to 2.0 mg over a 10 day period. After, participants continued on 2.0 mg daily for up to 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAF312 — BAF312 was provided as film-coated tablets in strengths of 0.25, 0,5, 1 and 2 mg for oral administration.
  Other Names: Siponimod
  Arms: BAF312 0.5mg; BAF312 10 mg; BAF312 2mg
Drug: Placebo — Matching placebo to BAF312 as tablets for oral administration.
  Arms: Placebo

SUMMARY:
This study investigated the dose response relationship for the efficacy and safety of BAF312 compared to placebo in active DM patients over a treatment period of 6+6 months and to determine the minimum dose required for a maximal clinical effect. The study was composed of 2 periods: a double-blind period 1 with BAF312 administered at different daily doses (0.5, 2, 10 mg and placebo) and a fixed-dose Period 2 in which BAF312 was administered at the dose of 2 mg daily .

DETAILED DESCRIPTION:
The study was prematurely terminated based on the results of an interim analysis where BAF312 did not demonstrate superior efficacy over placebo and a dose-response relationship was not observed. There were no safety concerns. Approximately 56 participants were planned to be randomized. A total of 17 participants were enrolled and randomized by the time the study was terminated.

ELIGIBILITY:
Key Inclusion Criteria:

Written informed consent must be obtained before any assessment is performed.

* Patients who have been defined as "definite" or "probable" based on the criteria of Bohan and Peter (Bohan and Peter 1975) for dermatomyositis at least 3 months before screening
* Patients must have active disease as defined by muscle weakness
* Patients may be on a stable dose of corticosteroid (up/equal to 20 mg once daily prednisone equivalent)
* Patients currently treated with oral or subcutaneous MTX must have been a stable dose of no more/equal to than 25 mg per week
* Patients currently treated with Azathioprine must have been a stable maintenance dose of no more/equal to 3 mg/kg/day
* Negative cancer screening conducted in the 12 months prior to screening visit

Key Exclusion Criteria

* Dermatomyositis patients having overlap myositis or any other type of myositis including paraneoplastic myositis, drug-induced myopathy, necrotizing myositis
* Preexisting severe cardiac or pulmonary conditions, malignancy of any organ system or significant eye diseases.
* Uncontrolled diabetes mellitus or diabetes complicated with organ involvement.
* Pregnant or nursing (lactating) women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-08-25 (Actual); Primary Completion 2016-02-17 (Actual); Study Completion 2016-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- United States (6):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, Boston, Massachusetts
- Novartis Investigative Site, Prague, Czech Republic, Czechia
- Japan (2):
  - Novartis Investigative Site, Chiba, Chiba
  - Novartis Investigative Site, Sendai, Miyagi

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=126

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was composed of 2 periods: a double-blind period 1 with BAF312 administered at different daily doses (0.5, 2, 10 mg and placebo) and a fixed-dose Period 2 in which BAF312 was administered to all randomized at the dose of 2 mg daily .
Pre-assignment Details: Participants were randomized to each treatment group in a1:1:1:1 ratio.
Period: Overall Study
Arm/Group | BAF312 0.5mg | BAF312 2mg | BAF312 10 mg | Placebo
Started | 5 | 4 | 4 | 4
Fixed Dose Period 2 | 5 | 4 | 4 | 4
Completed | 4 | 4 | 2 | 2
Not Completed | 1 | 0 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BAF312 0.5mg | BAF312 2mg | BAF312 10 mg | Placebo | Total
Number analyzed (Participants) | 5 | 4 | 4 | 4 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.8 (16.72) | 44.0 (6.98) | 51.8 (4.79) | 48.0 (10.61) | 49.1 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 4 | 3 | 13
  Male | 1 | 2 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Manual Muscle Testing - 24 Muscles (MMT-24) Score
Description: Each muscles tested was evaluated on a 0 - 10 scale where 0 indicated the weakest muscle score and 10 indicated the strongest muscle score. The total MMT24 score ranged from 0 - 240, where an increasing trend in the values indicates improvement. A positive change from baseline indicates improvement.
Time Frame: Baseline, 6 months
Population: The pharmacodynamic (PD) analysis set, which included all randomized participants, was considered for the analysis. Participants with valid baseline MMT24 score and at least one valid post baseline MMT24 score were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BAF312 0.5mg | BAF312 2mg | BAF312 10 mg | Placebo
Number analyzed (Participants) | 3 | 4 | 3 | 3
score on a scale | 28.286 (8.1539) | 12.367 (7.0967) | 14.026 (8.1541) | 27.735 (8.2175)
Statistical Analysis 1: Comparison: BAF312 0.5mg vs Placebo; Test type: Superiority or Other; p = 0.9621, Repeated measures analysis; Mean Difference (Net) = 0.551, 95% CI 2-sided [-22.447 to 23.549], Standard Error of Mean 11.5519
Statistical Analysis 2: Comparison: BAF312 2mg vs Placebo; Test type: Superiority or Other; p = 0.1637, Repeated measures analysis; Mean Difference (Net) = -15.368, 95% CI 2-sided [-37.128 to 6.391], Standard Error of Mean 10.9297
Statistical Analysis 3: Comparison: BAF312 10 mg vs Placebo; Test type: Superiority or Other; p = 0.2409, Repeated measures; Mean Difference (Net) = -13.709, 95% CI 2-sided [-36.806 to 9.388], Standard Error of Mean 11.6016

2. Secondary Outcome: BAF312 Plasma Concentration
Time Frame: 6 months
Population: Pharmacokinetics (PK) analysis set: The PK analysis set included all patients with available PK data and no protocol deviations with relevant impact on PK data.
Measure: Median (Full Range); unit: ng/ml
Arm/Group | BAF312 0.5mg | BAF312 2mg | BAF312 10 mg | Placebo
Number analyzed (Participants) | 3 | 4 | 2 | 0
ng/ml | 5.13 [3.96 to 6.31] | 25.9 [11.0 to 45.2] | 54.5 [50.9 to 58.0] |

3. Secondary Outcome: Peripheral Blood Lymphocyte Counts
Description: Absolute lymphocyte counts
Time Frame: baseline, 6 months
Population: Safety analysis set: the safety analysis set included all patients that received any study drug.
Measure: Mean (Standard Deviation); unit: 10^9 cells/Liter
Arm/Group | BAF312 0.5mg | BAF312 2mg | BAF312 10 mg | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 5
10^9 cells/Liter
  Baseline | 0.898 (0.3807) | 1.410 (0.7057) | 1.255 (0.6178) | 1.080 (0.0689)
  6 months: number analyzed (Participants) | 3 | 4 | 3 | 3
  6 months | 0.730 (0.4770) | 0.358 (0.0699) | 0.203 (0.0666) | 1.040 (0.190)

4. Secondary Outcome: Change From Baseline in Manual Muscle Testing - 24 Muscles (MMT-24) Score
Description: Each muscles tested was evaluated on a 0-10 scale where 0 indicated the weakest muscle score and 10 indicated the strongest muscle score. the total MMT24 score ranged from 0-240, where an increasing trend in the values indicates improvement. A positive change from baseline indicates improvement.
Time Frame: baseline, 3 months
Population: PD analysis set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | BAF312 0.5mg | BAF312 2mg | BAF312 10 mg | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4
score on a scale | 26.087 (7.0583) | 21.867 (7.0967) | 3.988 (7.0607) | 32.325 (7.1026)

5. Secondary Outcome: Change From Baseline in 6 Minutes Walking Distance (6-MWD) Test
Time Frame: baseline, 6 months
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | BAF312 0.5mg | BAF312 2mg | BAF312 10 mg | Placebo
Number analyzed (Participants) | 3 | 4 | 3 | 3
meters | 26.8 (104.15) | 22.2 (81.62) | 7.7 (66.73) | 4.1 (72.18)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 2.5 years
Groups:
- Period 1 Placebo: During period 1, participants received matching placebo daily for up to 24 weeks.
- Period 1 BAF312 0.5 mg/Day: During period 1, participants were uptitrated daily from BAF312 0.25 mg to 0.5 mg over a 10 day period. After, participants continued on 0.5 mg daily for up to 24 weeks.
- Period 1 BAF312 2 mg/Day: During period 1, participants were uptitrated daily from BAF312 0.25 mg to 2.0 mg over a 10 day period. After, participants continued on 2.0 mg daily for up to 24 weeks.
- Period 1 BAF312 10 mg/Day: During period 1, participants were uptitrated daily from BAF312 0.25 mg to 10.0 mg over a 10 day period. After, participants continued on 10.0 mg daily for up to 24 weeks.
- Period 2 Placebo /BAF312 2 mg/Day; Period 2 BAF312 0.5 mg/Day/BAF312 2 mg/Day; Period 2 BAF312 2 mg/Day/BAF312 2 mg/Day; Period 2 BAF312 10 mg/Day/BAF312 2 mg/Day: During period 2, participants were uptitrated daily from BAF312 0.25 mg to 2.0 mg over a 10 day period. After, participants continued on 2.0 mg daily for up to 24 weeks.
Arm/Group | Period 1 Placebo | Period 1 BAF312 0.5 mg/Day | Period 1 BAF312 2 mg/Day | Period 1 BAF312 10 mg/Day | Period 2 Placebo /BAF312 2 mg/Day | Period 2 BAF312 0.5 mg/Day/BAF312 2 mg/Day | Period 2 BAF312 2 mg/Day/BAF312 2 mg/Day | Period 2 BAF312 10 mg/Day/BAF312 2 mg/Day
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/4 | 0/4 | 1/4 | 0/5 | 0/4 | 1/4 | 1/4
Other Adverse Events (participants affected / at risk) | 1/5 | 1/4 | 4/4 | 4/4 | 2/5 | 1/4 | 4/4 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1 Placebo (N=5) | Period 1 BAF312 0.5 mg/Day (N=4) | Period 1 BAF312 2 mg/Day (N=4) | Period 1 BAF312 10 mg/Day (N=4) | Period 2 Placebo /BAF312 2 mg/Day (N=5) | Period 2 BAF312 0.5 mg/Day/BAF312 2 mg/Day (N=4) | Period 2 BAF312 2 mg/Day/BAF312 2 mg/Day (N=4) | Period 2 BAF312 10 mg/Day/BAF312 2 mg/Day (N=4)
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1 Placebo (N=5) | Period 1 BAF312 0.5 mg/Day (N=4) | Period 1 BAF312 2 mg/Day (N=4) | Period 1 BAF312 10 mg/Day (N=4) | Period 2 Placebo /BAF312 2 mg/Day (N=5) | Period 2 BAF312 0.5 mg/Day/BAF312 2 mg/Day (N=4) | Period 2 BAF312 2 mg/Day/BAF312 2 mg/Day (N=4) | Period 2 BAF312 10 mg/Day/BAF312 2 mg/Day (N=4)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chorioretinal atrophy (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Gingival recession (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis orbital (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dacryocystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Carbon monoxide diffusing capacity decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pulmonary function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Exertional headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transient global amnesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Internal limiting membrane peeling (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.